CLINICAL TRIAL: NCT05346393
Title: Hepatorenal Syndrome-acute Kidney Injury (HRS-AKI) Treatment With Transjugular Intrahepatic Portosystemic Shunt in Patients With Cirrhosis. A Randomized Controlled Trial
Brief Title: HRS-AKI Treatment With TIPS in Patients With Cirrhosis
Acronym: Liver-HERO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jena University Hospital (Other)
Collaborators: German Research Foundation (Other); University Hospital Halle (Saale) (Unknown)
Responsible Party: Principal Investigator, Cristina Ripoll, Prof. Dr., Jena University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZKSJ0146; DE-22-00013779 (Other: BfArM); 431667134 (Other Grant/Funding Number: DFG)
Record Dates: First submitted 2022-04-01; First posted 2022-04-26 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Cirrhosis, Liver; Hepatorenal Syndrome; Acute Kidney Injury; Ascites Hepatic
Keywords: Ascites; Acute Kidney Injury; Cirrhosis; Hepatorenal Syndrome; TIPS; transjugular intrahepatic portosystemic shunt; Terlipressin
MeSH Terms: conditions — Liver Cirrhosis; Hepatorenal Syndrome; Acute Kidney Injury; Ascites; Fibrosis | interventions — Portasystemic Shunt, Transjugular Intrahepatic; Standard of Care; Terlipressin; Albumins

STUDY DESIGN:
Intervention Model Description: Parallel Assignment 1:1-randomization, parallel design, stratified by center and AKI stage.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TIPS group (Experimental): TIPS implant (transjugular intrahepatic portosystemic shunt)
  Interventions: Procedure: TIPS
- Control group (Active Comparator): Standard medication therapy with terlipressin and albumin. In the case Terlipressin is not tolerated treatment with Noradrenaline may be considered following actual guidelines.
  Interventions: Drug: Standard of Care

INTERVENTIONS:
Procedure: TIPS — A transjugular intrahepatic portosystemic shunt (TIPS) is implanted into the cirrhotic liver
  Arms: TIPS group
Drug: Standard of Care — Terlipressin/Albumin treatment is the preferred standard of care treatment. In the case Terlipressin is not tolerated treatment with Noradrenaline may be considered following actual guidelines.
  Other Names: Terlipressin + Albumin
  Arms: Control group

SUMMARY:
The study compares the effectiveness and safety of TIPS implantation in patients with HRS-AKI (stage1, 2 and 3) and liver cirrhosis with standard therapy (drug therapy with terlipressin + albumin).

DETAILED DESCRIPTION:
Cirrhosis is a major cause of global health burden worldwide. Acute kidney injury (AKI) occurs in 20% of hospitalized patients with cirrhosis. Acute kidney injury is a relatively new definition of renal failure which takes into account the dynamic changes in serum creatinine. Among the causes of AKI, hepatorenal syndrome-AKI has the worst prognosis. HRS-AKI is an acute condition which occurs in patients with ascites, mainly refractory ascites. HRS-AKI includes the traditional hepatorenal syndrome type 1, which was defined by a serum creatinine cutoff and which has an ominous prognosis when left untreated, nevertheless HRS-AKI also includes milder forms of renal failure.

The standard treatment of HRS-AKI is with the infusion of albumin and terlipressin. Although this treatment improves renal function, patients remain at risk for new episodes of HRS-AKI and liver transplantation should be considered. Nevertheless, this optimal solution is only a reality for a privileged few given the shortage of organs and the common presence of contraindications.

Development of HRS-AKI is caused by increased pressure in the portal vein (the vein which brings the blood from the intestines to the liver), among other factors. Increased pressure in the portal vein, also called portal hypertension, is one of the main pathophysiological mechanisms that lead to the different complications of cirrhosis. Transjugular intrahepatic portosystemic shunt (TIPS) is an interventional radiological procedure which reduces the pressure in the portal vein by creating a short-cut between the portal vein and the hepatic vein, the vein which brings the blood from the liver towards the heart. TIPS placement has become the mainstay of treatment of some complications of cirrhosis, namely variceal bleeding and refractory ascites. Although rationally plausible, the use of TIPS in HRS-AKI has not been evaluated in the context of randomized controlled trials. Indirect data suggest that it could be helpful, since patients who become TIPS have an improvement in renal hemodynamics and renal function as well as less episodes of HRS-AKI in the follow-up. On the other hand, traditional HRS type 1 can be associated to liver failure and cardiac alterations which contraindicate TIPS placement. HRS-AKI includes not only traditional HRS type 1, but also milder forms of the disease, so that it is reasonable to consider that TIPS placement may have a role in this condition.

This study is a multicenter (14 centers), prospective, randomized controlled trial which evaluates use of TIPS in patients with HRS-AKI (stage 1, 2 and 3) versus standard of care (albumin and terlipressin). Patients with cirrhosis and HRS-AKI who fulfill the inclusion criteria and do not have any exclusion criteria will be randomized to standard of care or standard of care and TIPS. Patients will be followed for a minimum of 12 months until the end of the trial. The main end-point is to compare the survival at the end of follow-up among the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with cirrhosis confirmed by histology or liver stiffness or with unequivocal signs in ultrasound, endoscopy and/or blood tests
2. Clinically evident ascites due to portal hypertension
3. HRS-AKI
4. Age: ≥ 18 to ≤ 80 years old at the time of consent
5. ECOG < 4 prior to hospital admission
6. Subject has been informed of the nature of the study, is willing to comply with all required follow-up evaluations within the defined follow-up visit windows and has signed an Ethics Committee (EC) approved consent form.
7. Female subjects of childbearing potential have a negative pregnancy test ≤ 7 days before the procedure and are willing to use a reliable method of birth control for the duration of study participation. Female subjects will be exempted from this requirement in case they are sterile, infertile, or have been post-menopausal for at least 12 months (no menses). A contraceptive method with a pearl index below 1% is assumed to be effective.

Exclusion Criteria:

1. Recent or current use of nephrotoxic drugs (NSAIDS, Aminoglycosides or high-dosed iodinated contrast medium) in the previous 72 hours before AKI diagnosis
2. Improvement of renal function after 1 day of diuretic removal and plasma volume expansion with albumin 1-1.5 gr/kg
3. Uncontrolled shock within the last 48 hours prior to randomization
4. Patients with uncontrolled infection (defined by a 20 % increase in inflam-matory parameters (CRP, leucocytes or insufficient decrease of PMN in ascitic fluid < 25 % from baseline in the case of a SBP) despite 48 hours of antibiotic treatment.
5. Patients with cardiac cirrhosis as defined by the development of cirrhosis in a patient with chronic heart failure due to a primary cardiac disease (is-chemic cardiomyopathy, hypertensive cardiomyopathy, etc.)
6. Patients with contraindications to TIPS placement (e.g. Bilirubin > 85.5 µmol/L (≙ 5 mg/dL), recurrent hepatic encephalopathy, clinically relevant pulmonary hypertension, aortic stenosis)
7. Patients with cavernous portal vein thrombosis, splenic vein thrombosis or mesenteric vein thrombosis
8. Patients with clinically significant cardiac disease (NYHA ≥ II)
9. Patients with diastolic dysfunction grade 3.
10. Patients with a reduced systolic function with an ejection fraction ≤ 50 %
11. Patients with ACLF grade 3
12. Patients with creatinine value > 442 µmol/L (≙ 5 mg/dL)
13. Patients with an acute variceal bleeding at the time of screening who have indication for pre-emptive TIPS and/or terlipressin.
14. Patients with refractory ascites as defined by the International Ascites Club (< 800 gr weight loss over 4 days in patients on low salt diet and high dose diuretics (spironolactone 400 mg /day and furosemide * 160 mg /day), or lower dose of diuretics with complications secondary to the use of diuretics such as hyponatremia, renal failure, hepatic encephalopathy. *equivalent dose of torasemide 40 mg/day
15. Patients with hepatocellular carcinoma outside of the Milan criteria
16. Patients with hepatocellular carcinoma within the Milan criteria in whom the tumor is located in the puncture tract.
17. Patients with benign liver tumors (except regenerative nodules) which are located in the puncture tract.
18. Patients who already have a TIPS placed
19. Patients who already had a liver transplantation
20. Patients with other comorbidities that lead to an estimated life expectancy under 1 year.
21. Patients with respiratory insufficiency which requires mechanical ventila-tion
22. Patients with circulatory failure which requires administration of other vas-opressors (catecholamines)
23. Patients receiving renal replacement therapy
24. The subject is currently enrolled in another investigational device or drug trial.
25. Patients with pregnancy or lactation
26. Patients which are suspected to be incompliant for study participation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2022-11-29 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
12 month Liver transplant-free survival | 12 months after Baseline
  12 month Liver transplant-free survival

SECONDARY OUTCOMES:
3-month liver transplant free survival | 3 months after Baseline
  3-month liver transplant free survival
Number of patient which develop an indication for TIPS placement (variceal bleeding or refractory ascites) or TIPS revision (variceal bleeding or development of ascites) during follow-up | within 12 months after Baseline
  Number of patient which develop an indication for TIPS placement according to clinical guidelines (such as variceal bleeding or refractory ascites) in the control group or indication for a TIPS revision (variceal bleeding, development of ascites) in the intervention group will be assessed during the 12 months follow-up
Development of further decompensation of HRS-AKI during follow-up | within 12 months after Baseline
  Development of further decompensation as defined in the Baveno VII Consensus Workshop (e.g. overt hepatic encephalopathy, refractory or recurrent ascites, dilutional hyponatremia, new AKI-HRS, variceal bleeding) during follow-up
Reversal of HRS-AKI-AKI 3 MFU | 3 months after Baseline
  Reversal of HRS-AKI-AKI at 3 months (vs. baseline), defined as return of serum creatinine level within 0.3 mg/dl (26 mmol/L).
Reversal of HRS-AKI-AKI 12 MFU | 12 months after Baseline
  Reversal of HRS-AKI-AKI at 12 months (vs. baseline), defined as return of serum creatinine level within 0.3 mg/dl (26 mmol/L).
Partial response to treatment 3 MFU | 3 months after Baseline
  Partial response to treatment at 3 months (vs. baseline) defined as reduction of at least one AKI stage with decrease of serum creatinine to ≥ 0.3 mg/dl (26 mmol/L) above the baseline value.
Partial response to treatment 12 MFU | 12 months after Baseline
  Partial response to treatment at 12 months (vs. baseline) defined as reduction of at least one AKI stage with decrease of serum creatinine to ≥ 0.3 mg/dl (26 mmol/L) above the baseline value.
In-hospital survival | baseline until 12 months
  In-hospital survival of the patients (patients are hospitalized for diagnosis of HRS-AKI and start of treatment - due to poor diagnosis, patients may die during hospital stay)
28-day survival | baseline until day 28 after baseline
  28-day survival
90-day survival | baseline until day 90 after baseline
  90-day survival
Length of in-hospital-stay | baseline until 12 months
  Length of in-hospital-stay of the patients (patients are hospitalized for diagnosis of HRS-AKI and start of treatment)
Changes in HrQoL as measured by SF36 3 MFU | 3 months after Baseline
  Relative changes in Health-related Quality of Life as measured by SF36 at 3 months (vs. baseline)
Changes in HrQoL as measured by SF36 12 MFU | 12 months after Baseline
  Relative changes in Health-related Quality of Life as measured by SF36 at 12 months (vs. baseline)
Changes in HrQoL as measured by CLDQ 3 MFU | 3 months after Baseline
  Relative changes in Health-related Quality of Life as measured by CLDQ (Chronic Liver Disease Questionnaire) at 3 months (vs. baseline)
Changes in HrQoL as measured by CLDQ 12 MFU | 12 months after Baseline
  Relative changes in Health-related Quality of Life as measured by CLDQ (Chronic Liver Disease Questionnaire) at 12 months (vs. baseline)
Need for renal replacement therapy | 12 months after Baseline
  Need for renal replacement therapy within Follow-up
recurrence of HRS-AKI after treatment at 3 months | 3 months after Baseline
  recurrence of HRS-AKI after treatment at 3 months
recurrence of HRS-AKI after treatment at 12 months | 12 months after Baseline
  recurrence of HRS-AKI after treatment at 12 months
Safety Assessment | 12 months after Baseline
  Number of AEs and SAEs in each group with special attention on the development of acute on chronic liver failure and signs of heart failure.
Development of acute-on-chronic liver failure during follow-up | 12 months after Baseline
  Development of acute-on-chronic liver failure during follow-up
Impact of the presence of intrinsic nephropathy as assessed by cystatin C and UnGAL on outcomes (survival and reversal of AKI) | 12 months after Baseline
  Patients with clear intrinsic nephropathy will be excluded from the study, as the diagnosis of hepatorenal syndrome requires exclusion of intrinsic nephropathy. Nevertheless, patients with HRS may also have other conditions that may lead to a subclinical chronic nephropathy. This will be assessed with cystitis C and/or UnGAL and its association with survival and reversal of AKI. This is a secondary exploratory end-point

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Ripoll, Prof. Dr., Study Director — Jena University Hospital
Locations (14):
- Germany (14):
  - University Hospital RWTH Aachen, Aachen
  - Charité - Universitätsmedizin Berlin CVK, Berlin
  - University Hospital Dresden, Medical Clinic I, Gastroenterology, Dresden
  - Universitätsklinikum Essen (AöR), Essen
  - University Hospital Freiburg, Freiburg im Breisgau
  - University Hospital Halle, Halle
  - University Hospital Hamburg-Eppendorf, Hamburg
  - Medical University Hannover, Hanover
  - Jena University Hospital, Clinic for Inner Medicine IV, Jena
  - Klinikum Landshut AdöR der Stadt Landshut, Landshut
  - University Hospital Leipzig, Leipzig
  - RKH Clinic Ludwigsburg, Ludwigsburg
  - Ludwig-Maximilians-University, Klinikum Großhadern, Munich
  - University Hospital Münster, Medical Clinic B, Münster

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gonzalez-Garay AG, Serralde-Zuniga AE, Velasco Hidalgo L, Flores Garcia NC, Aguirre-Salgado MI. Transjugular intrahepatic portosystemic shunts for adults with hepatorenal syndrome. Cochrane Database Syst Rev. 2024 Jan 18;1(1):CD011039. doi: 10.1002/14651858.CD011039.pub2. PMID 38235907
- [Derived] Ripoll C, Platzer S, Franken P, Aschenbach R, Wienke A, Schuhmacher U, Teichgraber U, Stallmach A, Steighardt J, Zipprich A; Liver-HERO Study Group. Liver-HERO: hepatorenal syndrome-acute kidney injury (HRS-AKI) treatment with transjugular intrahepatic portosystemic shunt in patients with cirrhosis-a randomized controlled trial. Trials. 2023 Apr 5;24(1):258. doi: 10.1186/s13063-023-07261-9. PMID 37020315

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-03): https://cdn.clinicaltrials.gov/large-docs/93/NCT05346393/Prot_SAP_000.pdf